CLINICAL TRIAL: NCT06306924
Title: UNC Metastatic Cancer Radiation Therapy Registry
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2303
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Metastatic Cancer
Keywords: radiation therapy
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative radiation therapy: Subjects who are with metastatic cancer receive palliative radiation therapy.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Subjects with metastatic cancer receive radiation therapy.

SUMMARY:
The purpose of this registry is to collect clinical data from participants attending UNC Hospitals who present with metastatic cancer and are evaluated to receive radiation therapy as part of their standard of care treatment. The goal of this study is to provide a foundation for studies designed to identify projects across the translational continuum related to metastatic cancer and radiation therapy treatment. The relevant clinical data will be linked to patient-reported outcomes (PROs) thus allowing for a unique and robust dataset. Ultimately, this registry will provide current and future studies with the ability to analyze the correlation of radiation therapy regimens with metastatic cancer outcomes.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent was obtained to participate in the study and HIPAA

Authorization for release of personal health information. Ability to understand and willingness to sign informed consent

Diagnosed with or is suspected to have metastatic cancer.

Age ≥ 18 years at the time of consent.

Evaluated to receive radiation therapy as part of their standard-of-care treatment plan.

Exclusion Criteria:

All participants must not meet any of the following exclusion criteria prior to enrollment to participate in this study:

Any serious medical or psychiatric disorder that would interfere with the participant's ability to give informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with metastatic cancer receiving palliative radiation therapy at the University of North Carolina Chapel Hill.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-21 (Actual); Primary Completion 2033-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Data | Up to 1 month
  Clinical data and radiological assessments from participants with metastatic cancer receiving radiation therapy as a part of the standard of care will be collected.

SECONDARY OUTCOMES:
Patient reported outcomes (PRO) | Baseline, 1 month, 3 months, 6 months, 9 months, and 12 months
  Patient reported outcomes (PRO) from participants will be collected at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Sud, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials